CLINICAL TRIAL: NCT01448681
Title: A Continuous, Non-Invasive, Real-time Method for Estimating and Predicting Intracranial Hypertension
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 10-1412
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Intracranial Hypertension; Elevated ICP (Intracranial Pressure)
Keywords: Intracranial Hypertension; Elevated ICP (Intracranial Pressure)
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SICU patients with ICP: Surgical intensive care unit patients with elevated intracranial pressure
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions

SUMMARY:
There is statistically significant correlation between invasive measures of intracranial pressure (ICP) and non-invasive, real-time, continuous physiologic waveform data algorithms to predict ICP. Furthermore, characteristics within this physiologic waveform data will allow modeling for trend prediction of derived ICP information. Specific aims:

1. Develop models to estimate ICP and cerebral perfusion pressure (CPP) after traumatic brain injury in humans.
2. Predict and anticipate changes in ICP for preemptive management purposes.
3. Analyze characteristics of changes in ICP after treatment failure.
4. Analyze data to predict/anticipate confounding physiologic factors that affect ICP and its treatment.
5. Test the resulting models in real time.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe traumatic brain injury resulting in motor Glasgow Coma Score (GCS) score < 5
* age 18-89 years
* health care provider indicating the need for hyperosmolar therapy for elevated ICP

Exclusion Criteria:

* pregnancy
* incarceration
* brain death (GCS 3 with fixed, dilated pupils)
* life-threatening systemic injuries (Abbreviated Injury Scale (AIS) >4 in an organ system other than CNS)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Algorithm development | 24 months
  Developing algorithms relating data to intracranial pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Moulton, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States